CLINICAL TRIAL: NCT00722319
Title: Ongoing WARfarin and Coronary STENTing. A Multi-center, Prospective Registry on Antithrombotic Treatment.
Brief Title: Ongoing WARfarin and Coronary STENTing
Acronym: WAR-STENT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: War-Stent Investigators (Other)
Responsible Party: Aldo P. Maggioni, Associazione Nazionale Medici Cardiologi Ospedalieri (ANMCO)
Other Study IDs: WS-1
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2010-01

CONDITIONS: Acute Coronary Syndrome; Atrial Fibrillation
Keywords: oral anticoagulation; warfarin; percutaneous coronary intervention; stent; antiplatelet agents
MeSH Terms: conditions — Acute Coronary Syndrome; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients on long-term oral anticoagulation who are submitted to PCI-S because of acute coronary syndrome or stable angina. No further groups nor interventions are anticipated since the study is observational

SUMMARY:
Patients on warfarin treatment pose particular problems when undergoing percutaneous coronary intervention with stent implantation (PCI-S), because of the poor definition of the optimal antithrombotic strategies to be adopted both peri-procedurally and during the 4 (or more) weeks after PCI-S, when dual antiplatelet therapy with aspirin and clopidogrel is recommended. In the absence of solid evidence-based data, no definite recommendations for the management of this patient subset are currently given in the guidelines on percutaneous coronary intervention issued by the most prominent Cardiology Associations. Indeed, a high variability has been reported in the current antithrombotic strategies, which may consist in either the temporary substitution of warfarin by dual antiplatelet treatment or the combination of warfarin and aspirin or clopidogrel or both. Peri-procedural bridging therapy with either intravenous unfractionated or subcutaneous low-molecular-weight heparin is also variably carried out. Purpose of this registry is to determine in patients on warfarin treatment undergoing PCI-S: 1) the contemporary peri-procedural and medium-term antithrombotic management; and 2) the relative safety and efficacy of the various antithrombotic regimens.

DETAILED DESCRIPTION:
Patients on oral anticoagulation with vitamin-K antagonists who undergo PCI-S will be prospectively included in the registry and follow up for 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patients with ongoing warfarin treatment.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with warfarin who are hospitalized at tertiary centers all over the country to undergo percutaneous coronary intervention with stent implantation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of major/minor bleeding + adverse cardiac events (i.e., need for urgent re-revascularization, myocardial infarction, death) + arterial/venous thrombosis/thromboembolism | 1, 3, 6 and 12 months

SECONDARY OUTCOMES:
Incidence of major/minor bleeding | 1, 3, 6 and 12 months
Adverse cardiac events (i.e., need for urgent re-revascularization, myocardial infarction, death) | 1, 3, 6 and 12 months
Stent thrombosis | 1, 3, 6 and 12 months
Arterial/venous thromboembolism; | 1, 3, 6 and 12 months
Blood transfusions | 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rubboli, MD, Study Director — Division of Cardiology, Maggiore Hospital, Bologna
Locations (1):
- Division of Cardiology, Bologna, Italy

REFERENCES:
- [Background] Rubboli A, Halperin JL, Airaksinen KE, Buerke M, Eeckhout E, Freedman SB, Gershlick AH, Schlitt A, Tse HF, Verheugt FW, Lip GY. Antithrombotic therapy in patients treated with oral anticoagulation undergoing coronary artery stenting. An expert consensus document with focus on atrial fibrillation. Ann Med. 2008;40(6):428-36. doi: 10.1080/07853890802089786. PMID 18608125
- [Background] Rubboli A, Verheugt FW. Antithrombotic treatment for patients on oral anticoagulation undergoing coronary stenting: a review of the available evidence and practical suggestions for the clinician. Int J Cardiol. 2008 Jan 24;123(3):234-9. doi: 10.1016/j.ijcard.2007.02.017. Epub 2007 Apr 16. PMID 17434621
- [Background] Rubboli A, Colletta M, Herzfeld J, Sangiorgio P, Di Pasquale G. Periprocedural and medium-term antithrombotic strategies in patients with an indication for long-term anticoagulation undergoing coronary angiography and intervention. Coron Artery Dis. 2007 May;18(3):193-9. doi: 10.1097/MCA.0b013e328012a964. PMID 17429293
- [Background] Rubboli A, Di Pasquale G. The combination of anticoagulant and anti-platelet therapy in patients with atrial fibrillation: a comment on the recent ACC/AHA/ESC guidelines for the management of patients with atrial fibrillation. Eur Heart J. 2006 Dec;27(23):2908-9; author reply 2909-10. doi: 10.1093/eurheartj/ehl348. Epub 2006 Oct 30. No abstract available. PMID 17074773
- [Background] Rubboli A, Milandri M, Castelvetri C, Cosmi B. Meta-analysis of trials comparing oral anticoagulation and aspirin versus dual antiplatelet therapy after coronary stenting. Clues for the management of patients with an indication for long-term anticoagulation undergoing coronary stenting. Cardiology. 2005;104(2):101-6. doi: 10.1159/000086918. Epub 2005 Jul 12. PMID 16020950
- [Background] Rubboli A, Colletta M, Di Pasquale G. Regarding antithrombotic treatment after coronary stenting in patients on chronic oral anticoagulation. Am Heart J. 2005 Feb;149(2):E1. doi: 10.1016/j.ahj.2004.08.019. No abstract available. PMID 15846242
- [Derived] Rubboli A, Saia F, Sciahbasi A, Leone AM, Palmieri C, Bacchi-Reggiani ML, Calabro P, Bordoni B, Piccalo G, Franco N, Nicolino A, Magnavacchi P, Vignali L, Mameli S, Dallago M, Maggiolini S, Steffanon L, Piovaccari G, Di Pasquale G; WARfarin and Coronary STENTing (WAR-STENT) Study group. Twelve-month outcome of patients with an established indication for oral anticoagulation undergoing coronary artery stenting and stratified by the baseline risk of bleeding: Insights from the Warfarin and Coronary Stenting (War-Stent) Registry. Cardiovasc Revasc Med. 2017 Sep;18(6):425-430. doi: 10.1016/j.carrev.2017.03.015. Epub 2017 Mar 19. PMID 28363682
- [Derived] Rubboli A, Saia F, Sciahbasi A, Bacchi-Reggiani ML, Steffanon L, Briguori C, Calabro P, Palmieri C, Rizzi A, Imperadore F, Sangiorgi GM, Valgimigli M, Carosio G, Steffenino G, Galvani M, Di Pasquale G, La Vecchia L, Maggioni AP, Bolognese L; WARfarin and Coronary STENTing (WAR-STENT) Study Group. Outcome of patients on oral anticoagulation undergoing coronary artery stenting: data from discharge to 12 months in the Warfarin and Coronary Stenting (WAR-STENT) Registry. J Invasive Cardiol. 2014 Nov;26(11):563-9. PMID 25363997
- [Derived] Rubboli A, Sciahbasi A, Briguori C, Saia F, Palmieri C, Moroni LA, Calabro P, Leone AM, Franco N, Valgimigli M, Varani E, Santi M, Pasqualini P, Capecchi A, Piccalo G, Margheri M, di Pasquale G, Galvani M, Bolognese L, Gonzini L, Maggioni AP; WARfarin and coronary STENTing registry. In-hospital management and outcome of patients on warfarin undergoing coronary stent implantation: results of the multicenter, prospective WARfarin and coronary STENTing (WAR-STENT) registry. J Invasive Cardiol. 2013 Apr;25(4):170-6. PMID 23549489
- [Derived] Rubboli A, Bolognese L, Di Pasquale G, Galvani M, La Vecchia L, Maggioni AP. A prospective multicentre observational study on the management of patients on oral anticoagulation undergoing coronary artery stenting: rationale and design of the ongoing warfarin and coronary stenting (WAR-STENT) registry. J Cardiovasc Med (Hagerstown). 2009 Feb;10(2):200-3. doi: 10.2459/JCM.0b013e3283212f07. PMID 19377385